CLINICAL TRIAL: NCT06146400
Title: Role of CBC Parameters in Early Diagnosis of Bacterial and Viral Pediatric Pneumonia
Brief Title: Role of CBC Parameters in Early Diagnosis of Pediatric Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Abdeltwab saber, Principle investigator, Assiut University
Other Study IDs: pediatric pneumonia
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Infectious Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detection of the role of Complete Blood Count (CBC) parameters in early diagnosis of pediatric pneumonia

-Testing the ability of Complete Blood Count (CBC) parameters (N/L ratio, PLT /MPV ratio, MPV and other parameters) to differentiate between viral and bacterial pneumonia.

DETAILED DESCRIPTION:
Pneumonia is the leading cause of hospitalizations and death among children with nearly 120 million new cases and one million deaths every year.

* Viruses are the main cause of pneumonia in infants and toddlers between 30 days and 2 years old.
* Children 2 to 5 years old, respiratory viruses are also common with the rise of cases related to S. pneumoniae and H. influenzae type B and other bacterial organisms.

Viral pneumonia caused by , respiratory syncytial virus, which are the most common cause of community- acquired pneumonia in children younger than 5 years. Streptococcus pneumoniae is the most common bacterial cause across all age groups. Other important bacterial causes in children younger than 5 years include Hemophilus influenzae, Streptococcus pyogenes, Staphylococcus aureus, and Moraxella catarrhalis.

Parapneumonic effusion/empyema (PPE/EP), necrosis of lung parenchyma (NC), and lung abscess (AB), are serious complication of pediatric pneumonia. Because of these serious complications, early diagnosis of the causative organism is very important to start the proper treatment and avoid these serious complications.

Complete Blood Picture (CBC) is one of the most important preliminary routine investigations for diagnosis and monitoring of infection.

Recently, CBC parameters, especially Total Leucocyte Count (TLC), ANC, and platelet count all showed significant associations with neonatal sepsis. Besides, the TLC,Absolute neutrophils count (ANC), and platelet counts had good sensitivity and specificity in diagnosing neonatal sepsis

Another study have assessed the utility of C-reactive protein (CRP), White Cell Count (WCC), Neutrophil/Lymphocyte ratio (N/L), Platelets/ Mean Platelets Volume ratio (PLT/MPV ratio), Mean Platelets Volume (MPV), Monocyte Distribution Width (MDW) and many other CBC ratios to differentiate probable bacterial infections from non-bacterial infections and also assessed the severity of illness.

- In this study, we are going to test the role of Complete Blood Picture (CBC) parameters and ratios as an early detection tool of bacterial and viral pneumonia. This might have a role in early prediction and diagnosis of the causative organism. Which in turn leads to rapid intervention, and better prognosis.

ELIGIBILITY:
Inclusion Criteria:

-

Newly suspected cases of pneumonia from age o 1 month to 5 years in 2 age groups

Exclusion Criteria:

* Age group >5 years
* Already diagnosed patient who is under treatment

Ages: 1 Year to 5 Years | Sex: All
Age Groups: Child
Study Population: * Based on determining the main outcome variable, the estimated minimum required sample size is 80 suspected cases of pneumonia and 80 controls.
  * The sample size was calculated using Epi-info version 7 software, based on the following assumptions: Main outcome variable is the role of Complete Blood Count (CBC) parameters in early diagnosis of pediatric pneumonia. Based on previous studies (put reference) the percentage children of under 5 years who had pneumonia was 25.6% and based on the percentage confidence limits of 6% and a Confidence level =80%
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
role of CBC parameters and ratios in early diagnosis of pediatric pneumonia - Detecting the role of Complete Blood Picture parameters and ratios in early diagnosis of pediatric pneumonia CBC Parameters in diagnosis pediatric pneumonia | Baseline
  CBC parameters and ratios N/L Ratio PLT/MPV ratio ,MPV in differentiation between bacterial and viral pneumonia

IPD SHARING:
Plan to Share IPD: Undecided